CLINICAL TRIAL: NCT04353999
Title: The Effect of Diode Laser Photocoagulation on the Soft Tissue Healing During Socket Preservation in the Esthetic Zone.
Brief Title: The Effect of Laser Photocoagulation on the Soft Tissue Healing During Socket Preservation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ORG 0008839
Record Dates: First submitted 2020-04-11; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Soft Tissue Healing

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 980 nm diode laser photocoagulation (Experimental): 980 nm diode laser was used to coagulate the blood over the bone graft particles and achieve a socket seal after socket grafting
  Interventions: Procedure: Socket sealing by diode laser photocoagulation
- Dense polytetrafluroethylene membrane (Active Comparator): dPTFE membrane was used to seal the socket after grafting
  Interventions: Procedure: socket sealing with dense polytetrafluroethylene membrane

INTERVENTIONS:
Procedure: Socket sealing by diode laser photocoagulation — tooth extraction followed by socket grafting with bovine bone xenograft and finally sealed using 980 nm diode laser photocoagulation applied in a non-contact mode with a poer output of 1 watt in a continuous wave mode for 3-5 minutes
  Arms: 980 nm diode laser photocoagulation
Procedure: socket sealing with dense polytetrafluroethylene membrane — tooth extraction followed by socket grafting with bovine bone xenograft and finally sealed by a non-resorbable dPTFE membrane that is stabilized by suturing to the soft tissue margins of the socket
  Arms: Dense polytetrafluroethylene membrane

SUMMARY:
The main aim of this study was to evaluate clinically the effect of laser photocoagulation in comparison to the non-resorbable dense polytetrafluroethylene (dPTFE) membrane on the soft tissue healing during socket preservation with bovine bone xenograft.

DETAILED DESCRIPTION:
The study was designed as randomized, controlled, clinical trial. patients who were undergoing tooth extraction and socket preservation were divided into two groups: Group I:980 nm Diode laser was used to seal the socket by photocoagulation .Group II : a non-resorbable dPTFE was used to seal the socket and stabilized by suturing to the soft tissue margins of the socket

All patients were clinically and radiographically evaluated at the baseline and on the second , third and fourth weeks postoperatively.Then recalled after 4 months for the final radiographic examination.

ELIGIBILITY:
Inclusion Criteria:

1. The need for the extraction of nonrestorable maxillary anterior tooth for untreatable caries, endodontic treatment failure or root fracture.
2. Type I postextraction sockets according to the classification proposed by Elian et al. with all bony walls intact .
3. Adult patients (aged 18-50 years).
4. A good standard of oral hygiene, as determined by the registration of an O'Leary Plaque Index of less than or equal to 10% after phase I therapy.

Exclusion Criteria:

1. The presence of any systemic disease that could complicate bone and soft tissue healing of the grafted socket.
2. The presence of any local factor that may interfere with extraction as tooth ankylosis.
3. Smoking.
4. The presence of bone dehiscence and fenestrations of the post-extractive alveolus (Type II and III sockets).
5. Subjects who had undergone radiation therapy.
6. Patients who had been subjected to or who were under bisphosphonate therapy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Soft tissue healing (the changes in the soft tissue color throughout the first month) | at 2nd, 3rd and 4th week
  clinical examination and scoring according to Landry healing index. A score of 1 to 5 was given to the surgical site indicating the improvement of the nature of the soft tissue . A score of 1 meaning the least healing and 5 being excellent healing.

SECONDARY OUTCOMES:
soft tissue thickness in millimeters. | 4 months
  The thickness of the soft tissue in the center of the socket was measured at the baseline and after 4 months on the cone beam computed tomoghraph using the ruler tool to measure the thickness in millimeters.
Bone width and height measured in millimeters | 4 months
  bone dimensions were measured on the baseline cone beam computed tomograph and after 4 months also on the recall cone beam computed tomograph.
pain score on the visual analogue scale (VAS) | 1 week
  Pain was measured on the first , forth and seventh day postoperatively. The visual analogue scale comprises a scale graded from 1 to 100 to express the pain on a a ruler the the patient uses to point out the pain score visually with 0 meaning no pain and 100 meaning maximum pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A kamal, BDs, Principal Investigator — Alexandria University
Locations (1):
- Faculty of dentistry,Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Landry R, Turnbell R, Howley T. Effectiveness of benzydamyne HCl in the treatment of periodontal post-surgical patients. Res Clin Forums. 1988;10:105-118.
- [Background] Abrams L. Augmentation of the deformed residual edentulous ridge for fixed prosthesis. Compend Contin Educ Gen Dent. 1980 May-Jun;1(3):205-13. No abstract available. PMID 6950834
- [Background] Johnson K. A study of the dimensional changes occurring in the maxilla following tooth extraction. Aust Dent J. 1969 Aug;14(4):241-4. doi: 10.1111/j.1834-7819.1969.tb06001.x. No abstract available. PMID 5259350
- [Result] Schropp L, Wenzel A, Kostopoulos L, Karring T. Bone healing and soft tissue contour changes following single-tooth extraction: a clinical and radiographic 12-month prospective study. Int J Periodontics Restorative Dent. 2003 Aug;23(4):313-23. PMID 12956475